CLINICAL TRIAL: NCT02655107
Title: Non-invasive Measurement of Hemoglobin in Infants and Neonates: Comparison With CO-oximetrie and Point-of-care Devices.
Brief Title: Non-invasive Measurement of Hemoglobin in Infants and Neonates
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, PhD, University Hospital Schleswig-Holstein
Other Study IDs: AZ 119/14
Record Dates: First submitted 2015-12-05; First posted 2016-01-13 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Hemoglobins
Keywords: blood gas monitoring; non-invasive; hemoglobin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-invasive measurement of hemoglobin in infants and neonates scheduled for elective congenital heart surgery, weighing between 3kg and 20 kg. SpHb measurement will be compared to the gold standard of hemoglobin measurement - CO-oximetrie - and to the point-of-care (GEM 3500 premiere).

DETAILED DESCRIPTION:
Non-invasive measurement of hemoglobin in infants and neonates scheduled for elective congenital heart surgery, weighing between 3kg and 20 kg. SpHb measurement will be compared to the gold standard of hemoglobin measurement - CO-oximetrie - and to the point-of-care (GEM 3500 premiere). Data collection whenever an arterial blood gas analysis is indicated by the experienced attending anesthetist - before and after cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective congenital heart surgery
* routine use of an arterial line
* weight >= 3000g

Exclusion Criteria:

* urgent surgery
* premature birth
* parents refuse

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and neonates undergoing congenital heart surgery weighing between 3kg and 20kg
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin measurement non-invasively compared to gold standard hemoglobin | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Renner, PD Dr., Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No